CLINICAL TRIAL: NCT01205867
Title: An Open, Non-controlled, Non-randomised, Parallel-group Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of AZD 8848 Administered Intranasally to Male and Female Butyrylcholinesterase Deficient Subjects and to Sex and Age Matched Controls
Brief Title: Study to Investigate the Safety and Tolerability of AZD8848 in Butyrylcholinesterase Deficient Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0540C00009; EUDract No: 2010-019434-27
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Butyrylcholinesterase Deficiency
Keywords: Butyrylcholinesterase deficiency; tolerability; safety; AZD8848; pharmacokinetics; pharmacodynamics; BChE deficient subjects and matched control subject
MeSH Terms: conditions — Butyrylcholinesterase deficiency | interventions — AZD8848

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AZD8848 given to BChE deficient subjects and age & gender matched control subjects
  Interventions: Drug: AZD8848

INTERVENTIONS:
Drug: AZD8848 — Nasal spray solution, intranasal, single ascending doses, 1.4 - 60 μg

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of AZD8848 in Butyrylcholinesterase deficient subjects in comparison with sex and age matched control subjects.

DETAILED DESCRIPTION:
An Open, Non-controlled, Non-randomised, Parallel-group Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of AZD 8848 Administered Intranasally to Male and Female Butyrylcholinesterase deficient Subjects and to Sex and Age matched Controls

ELIGIBILITY:
Inclusion Criteria:

* BChE deficient subjects: The half-live of AZD8848 in plasma should be more than 20 minutes in an in vitro screening test
* Matched control subject: The half-live of AZD8848 in plasma should be less than 2 minutes in an in vitro screening test

Exclusion Criteria:

* Any clinically relevant abnormal findings in physical examination, laboratory assessments, vital signs or ECG
* Present or medical history of cardiovascular disease which, in the opinion of the investigator, may either put subject at risk because of participation in the study or influence the result of the study or the subject's ability to participate in the study
* Family history of autoimmune disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed by a panel of measurements including adverse events (AEs), vital signs, ECG, laboratory variables, physical examination, and clinical inspection of the nose | Immediately prior to administration of the IP (Day 0)
Safety and tolerability will be assessed by a panel of measurements including adverse events (AEs), vital signs, ECG, laboratory variables, physical examination, and clinical inspection of the nose | Repeated assessments during Day 1.
Safety and tolerability will be assessed by a panel of measurements including adverse events (AEs), vital signs, ECG, laboratory variables, physical examination, and clinical inspection of the nose | Repeated assessments during Day 2.

SECONDARY OUTCOMES:
Pharmacokinetics (concentration of AZD8848 and metabolite in plasma and urine) | Prior to administration of the IP (Day 0) and repeated assessments during the first 48h.
Pharmacodynamics (IL-1Ra in plasma) | Prior to administration of the IP (Day 0) and repeated assessments during the first 48h.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Sonne, MD, Principal Investigator — DanTrials ApS, Copenhagen, Denmark; Sam Lindgren, MD, PhD, Study Director — AstraZeneca R&D, Lund, Sweden
Locations (1):
- Research Site, Copenhagen, Copenhagen, Denmark

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1658&filename=D0540C00009_Study_Synopsis.PDF